CLINICAL TRIAL: NCT03424759
Title: An Open Label, Multicenter, Phase II Single-arm Trial of AZD9291 in Non-small Cell Lung Cancer (NSCLC) Patients With Uncommon Epidermal Growth Factor Receptor Mutations
Brief Title: Uncommon EGFR AZD9291
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Myung-Ju Ahn, Principal Investigator, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-06-176
Record Dates: First submitted 2018-01-09; First posted 2018-02-07 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AZD9291 (Experimental): Patients will be treated 80 mg/day of AZD9291 orally (1 cycle for 21 days).
  Interventions: Drug: AZD9291

INTERVENTIONS:
Drug: AZD9291 — Patients will be treated 80 mg/day of AZD9291 orally (1 cycle for 21 days).

SUMMARY:
EGFR (ErbB1) mutations define a lung cancer subtype with exquisite sensitivity to EGFR tyrosine kinase inhibitors (TKIs). While in-frame deletion in exon 19 (Del19) and a point mutation (L858R) in exon 21 are the two most common sensitizing EGFR mutations in NSCLC, approximately 10% of EGFR mutation-positive tumors harbor uncommon mutations.

These mutations represent a heterogeneous group of rare molecular alterations (or combinations) within exons 18-21, whose oncogenicity and sensitivity to EGFR TKIs may vary and has not been prospectively studied. Recently, a retrospective analysis reported that overall response rate of EGFR TKI (gefitinib or erlotinib) treatment was about 10% or less in Korean NSCLC patients with uncommon EGFR mutation other than del19, L858R and T790M [11]. In preclinical data, the potency of AZD9291 against uncommon EGFR mutants other than exon 20 insertion mutation was fairly good.

Based on the result, in this study, we try to evaluate the efficacy of AZD9291, the potent irreversible inhibitor, in NSCLC patients with harboring uncommon EGFR mutations.

DETAILED DESCRIPTION:
This is a single-arm phase II trial to evaluate the efficacy of AZD9291 (experimental) NSCLC patients with uncommon EGFR mutation. The primary endpoint of the study is objective response rate. Recently, a retrospective analysis reported that overall response rate of EGFR TKI (gefitinib or erlotinib) treatment was about 10% or less in Korean NSCLC patients with uncommon EGFR mutation other than del19, L858R and T790M (9).

In this study, we expect an objective response rate of about 30% for the experimental arm (AZD9291 therapy) compared to that of about 10% in the historical control based on previous studies. A sample size of 33 efficacy-evaluable patients would provide a power of 90% for testing the null hypothesis of 10% ORR vs. alternative hypothesis of 30% using a single-arm exact binomial test with a 1=sided significance level of 5%. The experimental therapy will be rejected if 6 or fewer patients out of 33 respond. Allowing for a follow-up loss rate of 10%, the total sample size is 37 patients.

Patients will be treated 80 mg/day of AZD9291 orally (1 cycle for 21 days). Subjects (with the exception of subjects with insulin dependent diabetes) must fast for ≥1 hours prior to taking a dose to ≥2 hour post dose. Water is permitted during this fasting period. Cycles were repeated until disease progression, unacceptable toxicity, or until the patient or the investigator requested therapy discontinuation. If the efficacy will be proven, the patient could receive the treatment continuously.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic or recurrent stage IV NSCLC with activating EGFR mutation other than deletion in exon 19, L858R, T790M and insertion in exon 20
* metastatic or recurrent NSCLC
* Be 19years of age on day of signing informed consent
* ECOG performance status of 0 to 2
* At least one measurable lesion by RECIST 1.1(The part of radiation treatment in the palliative setting is excluded.)
* Untreated asymptomatic brain metastasis or symptomatic brain metastasis treated with local treatment such as operation, whole brain radiotherapy, or gamma-knife surgery
* At least 2 weeks later after whole brain radiotherapy or at least 4 weeks later after palliative thoracic radiotherapy
* Adequate organ function as evidenced by the following; Absolute neutrophil count > 1.5 x 109/L; Hb > 9.0g/dL; platelets > 100 x 109/L; total bilirubin ≤1.5 UNL; AST and/or ALT < 2.5 ULN if no demonstrable liver metastases or < 5 UNL in the presence of liver metastases, CCr ≥ 50mL/min
* Written informed consent form

Exclusion Criteria:

* Prior treatment with EGFR TKI
* Major surgery undertaken less than 4 weeks before the study
* Localized palliative radiotherapy unless completed more than 2 weeks before the study
* Uncontrolled systemic illness such as DM, CHF, unstable angina, hypertension or arrhythmia
* Pregnant or nursing women (Women of reproductive potential have to agree to use an adequate contraceptive method)
* Uncontrolled symptomatic brain metastasis
* Prior history of malignancy within 5 years from study entry except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer, or well-treated thyroid cancer
* Concomitant use of CYP3A4 inducers/inhibitors
* Prolonged QT interval in ECG (QTc >450 msec)
* Prior history of interstitial lung disease

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | through study completion, an average of 2 years
  30%

CONTACTS AND LOCATIONS:
Overall Officials: Myung-Ju Ahn, Principal Investigator — Samsung Medical Center
Locations (1):
- Department of Medicine, Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cho JH, Lim SH, An HJ, Kim KH, Park KU, Kang EJ, Choi YH, Ahn MS, Lee MH, Sun JM, Lee SH, Ahn JS, Park K, Ahn MJ. Osimertinib for Patients With Non-Small-Cell Lung Cancer Harboring Uncommon EGFR Mutations: A Multicenter, Open-Label, Phase II Trial (KCSG-LU15-09). J Clin Oncol. 2020 Feb 10;38(5):488-495. doi: 10.1200/JCO.19.00931. Epub 2019 Dec 11. PMID 31825714